CLINICAL TRIAL: NCT04413266
Title: Effects of Curcumin Supplementation on Inflammation, Oxidative Stress and Microbiota in Patients With Chronic Kidney Disease on Peritoneal Dialysis
Brief Title: Effects of Curcumin Supplementation in Patients With Chronic Kidney Disease on Peritoneal Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Denise Mafra7
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Chronic Kidney Diseases; Peritoneal Dialysis; Hemodialysis
Keywords: chronic kidney disease; peritoneal dialysis; curcumin; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curcumin for CKD (Active Comparator): Administration of 3 capsules with 500mg of curcumin and piperine per day, for 12 weeks
  Interventions: Dietary Supplement: Curcumin supplementation
- Placebo for CKD (Placebo Comparator): Administration of 3 capsules with 500mg of placebo (maize starch) per day, for 12 weeks
  Interventions: Dietary Supplement: Curcumin supplementation

INTERVENTIONS:
Dietary Supplement: Curcumin supplementation — The patients will receive 3 capsules per day containing 500mg of curcumin for 4 weeks
  Other Names: Dietary Supplement; Placebo

SUMMARY:
The objective of this study is to assess whether supplementation with curcumin could modulate the intestinal microbiota, reducing levels of inflammatory markers of oxidative stress, uremic toxins and inflammasome, in patients with chronic kidney disease in peritoneal dialysis.

DETAILED DESCRIPTION:
Curcumin is a chemical compound of the curcuminoids class found in the root of Curcuma (Curcuma longa), and due to its potential antioxidant and anti-inflammatory, has been suggested as a nutritional strategy to reduce oxidative stress and inflammation present in several chronic diseases. Although it is a promising therapy, there are no studies evaluating the effects of curcumin in patients with chronic kidney disease (CKD) in peritoneal dialysis (PD). The aim of this study is to evaluate the effect of curcumin supplementation on inflammatory markers and oxidative stress in patients with CKD in PD. Methods: This is a longitudinal randomized clinical double-blind crossover study, with a washout period and placebo-controlled, where patients will be randomized into two groups: Turmeric and Placebo. After the 12-week supplementation period, a washout (12 weeks) will be performed for subsequent crossover of the patients. Mononuclear cells will be extracted from whole blood and the expression of m ribonucleic acid from transcription factors (Nrf2 and NF-kB), antioxidant enzymes (NQO1, HO-1), as well as NLRP3 inflammasome will be analyzed by real-time Polymerase Chain Reaction and protein expression by western blotting. Inflammatory cytokine levels will be assessed by ELISA, also, plasma levels of TBARS, routine laboratory parameters, as well as food intake and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Kidney Disease
* Peritoneal dialysis patients for more than 6 months
* Aged from 18 to 60 years
* Must be able to swallow tablets

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Using antioxidant supplements in the last 3 months
* Usual intake of turmeric
* Usual intake Autoimmune
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Antioxidants and anti-inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers- nuclear receptor factor 2 (Nrf2), glutathione peroxidase (GPx), heme oxygenase-1 (HO-1)
Inflammatory biomarkers | 4 weeks
  Get blood samples to evaluate the supplementation effects in inflammatory biomarkers- factor nuclear kappaB, interleukin 6 (IL-6), tumor necrosis factor-alpha (TNF-alpha), PCR, IL-18, TBARS, Inflammasome.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, Ph.D, Principal Investigator — Federal University Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Reis DCMV, Alvarenga L, Cardozo LFMF, Baptista BG, Fanton S, Paiva BR, Ribeiro-Alves M, Fortunato RS, Vasconcelos AL, Nakao LS, Sanz CL, Berretta AA, Leite M Jr, Mafra D. Can curcumin supplementation break the vicious cycle of inflammation, oxidative stress, and uremia in patients undergoing peritoneal dialysis? Clin Nutr ESPEN. 2024 Feb;59:96-106. doi: 10.1016/j.clnesp.2023.11.015. Epub 2023 Nov 28. PMID 38220413